CLINICAL TRIAL: NCT02291354
Title: A Randomized, Controlled Study of Synergism of Soluble Dietary Fiber With Fecal Microbiota Transplantation in Adult Patients With Slow Transit Constipation
Brief Title: Evaluating the Synergism of Soluble Dietary Fiber With Fecal Microbiota Transplantation in Slow Transit Constipation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIGS-Pectin-STC-2015
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-11

CONDITIONS: Slow Transit Constipation
Keywords: Fecal Microbiota Transplantation; Soluble Dietary Fiber; Slow Transit Constipation
MeSH Terms: interventions — Pectins; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT + Placebo (Placebo Comparator): Patients allocated to control group will receive standard FMT, followed by placebo for 12 weeks.
  Interventions: Other: Placebo; Procedure: Fecal microbiota transplantation (FMT)
- FMT + Pectin (Experimental): Patients allocated to experiment group will receive standard FMT, followed by 24g pectin each day for 12 weeks.
  Interventions: Drug: Pectin; Procedure: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Drug: Pectin — Patients allocated to experiment group will receive 12 g pectin each day for 12 weeks.
  Other Names: soluble dietary fiber
  Arms: FMT + Pectin
Other: Placebo — Patients allocated to experiment group will receive 12 g maltodextrin each day for 12 weeks.
  Arms: FMT + Placebo
Procedure: Fecal microbiota transplantation (FMT) — Standardized Frozen Fecal Microbiota will be infused via nasointestinal tube.
  Other Names: Fecal bacteriotherapy

SUMMARY:
The purpose of this study is to evaluate the synergism of Soluble Dietary Fiber with Fecal Microbiota Transplantation in Adult Patients with Slow Transit Constipation.

DETAILED DESCRIPTION:
Constipation is a chronic disease estimated to affect about 10% - 15% of the worldwide general population. Recent evidence in the literature and collected in our laboratory confirm that constipation can be a consequence of intestinal dysbiosis, which may affect the motility and metabolic environment of colon.

Fecal Microbiota Transplantation (FMT) is temporarily effective for patients with slow transit constipation. However, the transplanted microflora cannot maintain for a long time. Along with the gut microbiota returning to the original state, the symptoms relapse.

Pectin is a kind of soluble dietary fiber, producing short chain fatty acids (SCFAs) after a series of fermentation by gut flora to supply the energy for epithelial cells, regulate intestinal PH, promote intestinal motility and join effort in immune regulation with intestinal lymphoid tissue. Therefore, we conceive that pectin could promote the colonization of probiotics and reduce adhesion of pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Chronic constipation according to Rome III criteria, defined as two or fewer spontaneous, complete bowel movements (SCBMs) per week for a minimum of 6 months;
* Age ≥ 18 years;
* BMI: 18.5-25 kg/m2;
* Slow colonic transit confirmed by colonic transit test (colonic transit time (CTT) > 48 hours);
* Normal anorectal manometry, with no evidence of dyssynergia and confirmed ability to expel rectal balloon;
* No radiographic evidence of functional (i.e. pelvic floor dyssynergia) or anatomical (i.e. significant rectocele and intussusception) impediment to the expulsion of the radio-opaque contrast;
* Disease duration > 1 year;
* Traditional treatment with dietary modification, laxatives (including osmotic and stimulant laxatives), and biofeedback tried over the past 6 months without success;

Exclusion Criteria:

* Bowel constipation due to innate factor (i.e. megacolon) or secondary interventions (i.e. drugs, endocrine, metabolic, neurologic or psychologic disorders);
* History or evidence of gastrointestinal diseases (i.e. obstruction, cancer, inflammatory bowel diseases) ;
* Previous abdominal surgery, except cholecystectomy, appendicectomy, tubal ligation and cesarean section;
* Previous proctological or perianal surgery;
* A constipation condition meeting the Rome III criteria for IBS or functional abdominal pain syndrome;
* Pregnant or breast-feeding women;
* Infection with enteric pathogen;
* Usage of probiotics, prebiotics and/or synbiotics within the last month;
* Usage of antibiotics and/or PPIs within the last 3 months;
* Smoking or alcohol addiction within the last 3 months;
* Uncontrolled hepatic, renal, cardiovascular, respiratory or psychiatric disease;
* Disease or therapy with drugs (i.e. antidepressants, opioid narcotic analgesics, anticholinergics, calcium antagonists, nitrates, antimuscarinics) that, in the opinion of the investigator, could affect intestinal transit and microbiota.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having on average three or more SCBMs/week | 12 weeks
  Proportion of patients having on average three or more spontaneous, complete bowel movements (SCBMs) per week was evaluated at week 4 and 12.

SECONDARY OUTCOMES:
Bowel habit assessments | 12 weeks
  Patients kept daily diaries about times of bowel movements each day, stool consistency, degree of straining severity during defecation, and degree of sensation of incompleteness of evacuation.
Constipation-related symptoms assessments | 12 weeks
  Constipation-related symptoms were evaluated using the validated Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire at week 4 and 12.
Quality-of-Life assessments | 12 weeks
  Quality-of-Life was evaluated using the validated Patient Assessment of Constipation Quality of Life (PACQOL) self-report questionnaire at week 4 and 12.
Colonic transit time measurements | 12 weeks
  Colonic transit time (CTT) was measured at week 4 and 12 with the Metcalf method.
Usage of laxatives or enemas as rescue medication | 12 weeks
  If patients did not have a bowel movement for 3 or more consecutive days, they were permitted to take up to 20 g of Macrogol 4000 powder (Forlax). If ineffective, enema were used. Patients kept daily diaries about the rescue medication when used.
Adverse events | 12 weeks
  Adverse events include fever, diarrhea, abdominal pain, increased bloating, borborygmi, flatulence, nausea, vomiting, nasopharyngitis, and any other disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Study Director — Department of Generay Surgery, Jinling hosptal
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China